CLINICAL TRIAL: NCT00739778
Title: Effect of a Novel Sweetener on the pH of Dental Plaque.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cargill (Industry)
Responsible Party: Max Goodson, DDS, PhD, The Forsyth Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CFIS-08-001
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: food - novel sweetener — concentration to be isosweet with 4.7% sucrose
Other: food vehicle blank — water blank
Other: food - sweetener, positive control — 4.7% sucrose in water
Other: food - sweetener, negative control — non-cariogenic sweetener at concentration isosweet with 4.7% sucrose

SUMMARY:
Bacteria that live in the mouth can digest fermentable carbohydrates such as sucrose, fructose, and glucose to make acid. This acid can cause demineralization of the tooth and lead to dental caries or decay. Noncariogenic carbohydrate sweeteners, such as sugar alcohols, can be used to replace fermentable carbohydrates in foods, thereby decreasing the risk of caries. In order for a sweetener to be labeled as a noncariogenic sweetener, the FDA requires that when present in food, the food should not lower the dental plaque pH below 5.7 either during or up to 30 minutes after consumption. The purpose of this study is to determine whether a new developmental sweetener can be fermented by the bacteria in the mouth and lead to acid production. This will be done by measuring the pH of dental plaque following consumption of the sweetener.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as evidenced by the medical history.
* Male or non-pregnant, non-lactating females ages 18 to 75 inclusive.
* Caries experience in the past year.
* More than 5 decayed, missing, or filled teeth demonstrating a high caries experience.
* Acidogenic plaque as demonstrated by a drop in pH to 5.7 or lower when challenged with sucrose rinse at the screening visit.
* Willing to abstain from all oral hygiene procedures, brushing and flossing, for 48 hours prior to each test day and drink only water for the four (4) hours prior to each test.
* Willing to abstain from the use of mouthwashes during the study.

Exclusion Criteria:

* Presence of orthodontic appliances.
* Systemic conditions which could influence the pH of the oral cavity (i.e., diabetes, salivary gland disorders etc.).
* Use of medications that would influence the pH of the oral cavity. Specifically, concomitant use of neuroleptics, atropine, chemotherapeutic agents, diuretics, antibiotics, antihistamines, decongestants, and muscle relaxants. Also, anticipated need for intermittent use of any medications in these classes or history of use during the 72 hours immediately prior to the screening visit.
* Patients with aggressive periodontitis, acute necrotizing ulcerative gingivitis, or gross decay at discretion of Investigator.
* Females who by self report are pregnant, lactating, planning to be pregnant during the study period, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception during the study period.
* Exposure to any investigational agent within the 30 days prior to study visit 1
* Individuals requiring prophylactic antibiotics
* Allergy or intolerance to food ingredients and products including artificial sweeteners.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mean minimum plaque pH during the test period | 0-60 minutes

SECONDARY OUTCOMES:
Mean area under the pH-versus-time curve (AUC) | 0-60 min

CONTACTS AND LOCATIONS:
Overall Officials: Max Goodson, DDS, PhD, Principal Investigator — The Forsyth Institute
Locations (1):
- The Forsyth Institute, Boston, Massachusetts, United States